CLINICAL TRIAL: NCT04989179
Title: Incidence and Factors Affecting the Development and Outcome of Post Mastectomy Pain Syndrome - A Multi-centre Prospective Cohort Study.
Brief Title: Incidence and Factors Affecting the Development and Outcome of Post Mastectomy Pain Syndrome
Acronym: PMPS
Status: Active, not recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMPS 1
Record Dates: First submitted 2021-07-07; First posted 2021-08-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Post-mastectomy Pain Syndrome
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multi-centre, prospective study aims to obtain a precise estimate of the local incidence of PMPS and identify biopsychosocial risk factors contributing to the development of PMPS. Recognition of the impact of PMPS on function and mood and quality of life in cancer survivors, and identification of risk factors would help physicians institute appropriate pre-operative counselling and preventive measures to reduce the development of PMPS. The investigators aim to follow up on the long-term multi-dimensional effects of PMPS, and continue to develop and validate a risk prediction model for patients at risk of PMPS in the next phase of the study.

DETAILED DESCRIPTION:
Post-mastectomy pain syndrome (PMPS) has been reported to occur in 25-60% of patients following surgeries for breast cancer, the highest occurring cancer in women worldwide. There is a lack of an accepted standard definition of PMPS which has resulted in the wide range of estimates of its occurrence. While there has been much research interest in this condition, there is still a paucity of standardized and effective treatment at this point, and our understanding of this condition, its exact incidence and risk factors, is still incomplete.

The local incidence of PMPS after breast cancer surgery is presently unknown and often under-reported, although breast cancer surgery is common and is carried out in almost all Singhealth institutions. Risk factors for PMPS in the local context may differ from that postulated in the West due to cultural, racial and societal differences. Breast cancer has a high survival rate, with data from the CONCORD-2 study showing a 5-year survival rate of ≥85% in developed countries. Despite high survival rates in cancer survivors, PMPS has been shown to have a negative impact on the quality of recovery (QoR), patient satisfaction, and can be severe enough causing the diminished quality of life (QoL) including poor sleep, long-term disability, mood disorders and interference with activities of daily living (ADL).

Despite widespread recognition of PMPS, it is often untreated or undertreated. Some possible reasons suggested for inadequate management of PMPS are the lack of quality information about optimal treatment, and incomplete understanding of the mechanisms and risk factors for chronic pain development and prognosis. There is a knowledge gap in the understanding of risk factors leading to PMPS, the lack of a validated risk prediction model for development of PMPS, and hence limiting the institution of preventive analgesia in high risk patients. It is therefore timely to conduct a local multi-centre, prospective study to look at the local incidence of PMPS after breast surgery, the multi-dimensional effects of PMPS on the patient as well as to identify modifiable biopsychosocial risk factors leading to PMPS.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years old
* Provided consent for the study
* Types of breast surgery included: single or bilateral site mastectomies, with or without axillary clearance, wide excision with axillary clearance, radical mastectomies with or without flap surgery.

Exclusion Criteria:

1. Age below 21 or above 80 years old
2. Male patients
3. Cognitive impairment/ uncommunicative patients.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients will be recruited as breast cancer in male is very rare.
Study Population: Surgeons at the breast clinic listing patients for surgery will inform patients of the study. The clinical research coordinators will approach the potential study participants referred by the study team members and other attending pain clinicians.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Precise estimate of the local incidence and clinical/functional impact of PMPS | 4 months
  Hypothesized to result from damage to major peripheral nerves during surgery. The International Association for the Study of Pain (IASP) defines PMPS as persistent pain soon after mastectomy/lumpectomy affecting the anterior thorax, axilla, and/or medial upper arm. The primary outcome will be the local incidence of PMPS at 4 months follow-up after surgery.

SECONDARY OUTCOMES:
Identify risk factors of PMPS | 4 months
  Describe patient, anaesthetic and surgical factors (both modifiable and unmodifiable) contributing to the development of PMPS.
Describe factors likely to prevent or reduce the development of PMPS after breast cancer surgery | 4 months
  Identified risk factors can help to identify patients at risk of developing PMPS which then allows clinicians to institute prevention measures such as pre-operative counselling and preventive analgesics for high-risk patients with multiple risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Diana Chan, Principal Investigator — Singapore General Hospital
Locations (3):
- Singapore (3):
  - Singapore General hospital, Singapore, Singapore
  - Changi General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsson IM, Ahm Sorensen J, Bille C. The Post-mastectomy Pain Syndrome-A Systematic Review of the Treatment Modalities. Breast J. 2017 May;23(3):338-343. doi: 10.1111/tbj.12739. Epub 2017 Jan 30. PMID 28133848
- [Result] Small DM. Lateral chain packing in lipids and membranes. J Lipid Res. 1984 Dec 15;25(13):1490-500. PMID 6530598